CLINICAL TRIAL: NCT03760588
Title: PRevention of cArdiac Dysfunction During Adjuvant Breast Cancer Therapy: A Randomized, Placebo-controlled, Multicenter Trial
Brief Title: Prevention of Cardiac Dysfunction During Breast Cancer Therapy
Acronym: PRADAII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Torbjorn Omland (Other)
Collaborators: University Hospital, Akershus (Other); Oslo University Hospital (Other); University Hospital of North Norway (Other); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); Klinbeforsk (Other); Norwegian Cancer Society (Other); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Torbjorn Omland, Professor, University Hospital, Akershus
Organization: University Hospital, Akershus (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-004909-41
Record Dates: First submitted 2018-11-12; First posted 2018-11-30 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Female; Heart Failure
Keywords: LCZ696; CMR; Echocardiography; Cardio-oncology; Circulating biomarkers; Breast Cancer; Anthracyclines
MeSH Terms: conditions — Heart Failure; Breast Neoplasms | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, double blind design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril/valsartan (Experimental): Sacubitril/valsartan (target dose 97/103 mg b.i.d.) and matching placebo will be provided orally in a 1:1 parallel fashion stratified by study site and for planned treatment with trastuzumab. Dose titration will be performed as follows: Sacubitril/valsartan 24/26 mg b.i.d. will be administered for 2-4 weeks and provided blood pressure > 100 mmHg, no symptoms of hypotension or other side effects or adverse events (AE), followed by sacubitril/valsartan 49/51 mg b.i.d. for 2-4 weeks. Provided blood pressure > 100 mmHg, no symptoms of hypotension or other side effects or AE a further uptitration to sacubitril/valsartan 97/103 mg b.i.d. will be performed.
  Interventions: Drug: Sacubitril/valsartan
- Placebo (Placebo Comparator): Matched to the comparator.
  Interventions: Drug: Sacubitril/valsartan

INTERVENTIONS:
Drug: Sacubitril/valsartan — Target dose 97/103 mg b.i.d .
  Other Names: Entresto®

SUMMARY:
Breast cancer is the most common cancer among women. The modern post-surgery treatment with chemotherapy, immunotherapy, radiation and hormone therapy has improved the overall 5-years survival drastically. However, an unwanted effect of the post-surgery treatment is its potentially deleterious effect on the heart resulting in cardiac dysfunction. Angiotensin antagonists are used as part of the heart failure treatment. In smaller studies angiotensin antagonists have shown to have a cardioprotective effect during breast cancer treatment. Sacubitril/valsartan is a potent drug that in addition to an angiotensin antagonist contains a neprilysin inhibitor. Sacubitril/valsartan has proved to be superior to enalapril in chronic heart failure. In this randomized placebo controlled double blind trial we hypothesize that sacubitril/valsartan used concomitantly during anthracycline containing chemotherapy for breast cancer treatment prevents cardiac dysfunction as measured by cardiac magnetic resonance imaging (CMR). PRADA II is a Norwegian multicenter trial intending to recruit 214 patients and follow them for 18 months with CMR, cardiac ultrasound, blood samples, functional capacity tests and health related quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women with histological evidence of invasive early breast cancer scheduled for adjuvant therapy with anti-cancer regimens that include anthracyclines
* Eastern Cooperative Oncology Group performance status 0-1
* Sinus rhythm

Exclusion criteria:

* Age <18 years
* Renal failure, i.e. serum creatinine greater than 133 mol/L (1.5mg/dL) or estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73m2
* Hyperkalemia, i.e. serum potassium greater than 5.0 mmol/L
* Systolic blood pressure < 100 mgHg
* Uncontrolled hypertension
* Acute myocardial infarction within the last three months
* Contraindication to ACEI or ARB or sacubitril/valsartan, including previous hypersensitivity reaction, angioedema and renal artery stenosis
* ACEI, ARB, aldosterone antagonist or sacubitril/valsartan use within 4 weeks of study start
* Clear indication for ACEI, ARB, aldosterone antagonist or sacubitril/valsartan therapy, including symptomatic heart failure
* History of hemodynamically significant valvular disease
* Active liver disease, i.e. alanine aminotransferase or aspartate aminotransferase greater than 1.5 times the upper limit of normal
* Participation in another pharmaceutical clinical trial of an investigational medicinal product (IMP) less than 4 weeks prior to inclusion or use of other investigational drugs within 5 halflives of enrollment, whichever is longer
* Conditions that would affect the participants to comply with the study protocol as psychiatric or mental disorders, alcohol abuse or other substance abuse, suspected poor drug compliance, language barriers or other factors
* Contraindication or inability to undergo CMR examination
* Fertile women with inadequate birth control, pregnancy, and/or breastfeeding. Adequate contraception includes oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device or system, vasectomized partner or sexual abstinence. Fertile women are defined as following menarche and until becoming postmenopausal unless permanently sterile. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause
* Life expectancy < 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction by cardiovascular magnetic resonance | From randomization to end of blinded therapy (18 months)

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction by echocardiography | From randomization to end of blinded therapy (18 months)
Change in left ventricular systolic global longitudinal strain by echocardiography | From randomization to end of blinded therapy (18 months)
Change in left ventricular systolic global longitudinal strain by cardiovascular magnetic resonance (CMR) | From randomization to end of blinded therapy (18 months)
Change in left ventricular end-systolic volume measured by CMR | From randomization to end of blinded therapy (18 months)
Incidence of a significant reduction in left ventricular systolic function measured by CMR or echocardiography | From randomization to end of blinded therapy (18 months)
  An absolute reduction in LVEF ≥ 5% by CMR or a relative percentage reduction of global longitudinal strain (GLS) > 15%
Incidence of cardiotoxicity measured by CMR or echocardiography | From randomization to end of blinded therapy (18 months)
  Absolute reduction in LVEF ≥ 10% to a value below 50% as measured either by CMR or Echocardiography, or incidence of clinical heart failure
Change in circulating cardiac biomarkers | From randomization to end of blinded therapy (18 months)
  Cardiac biomarkers defined as cardiac troponins I and T measured by high sensitivity assays (hs-TnI and hs-TnT) and N-terminal proB-type natriuretic peptide (NT-proBNP)

OTHER OUTCOMES:
Incidence of adverse events and serious adverse events | From randomization to end of blinded therapy (18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Torbjørn Omland, MD,PhD,MPH, Principal Investigator — University Hospital, Akershus
Locations (4):
- Norway (4):
  - Akershus University Hospital, Lørenskog
  - Stavanger University Hospital, Stavanger
  - University of North Norway, Tromsø
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omland T, Heck SL, Holte E, Lilleaasen AM, Gynnild MN, Fagerland MW, Vinje-Jakobsen V, Naes AL, Blix ES, Larsen AI, Geisler J, Gulati G, Wethal T. Sacubitril/Valsartan and Prevention of Cardiac Dysfunction During Adjuvant Breast Cancer Therapy: The PRADA II Randomized Clinical Trial. Circulation. 2025 Oct 21;152(16):1136-1145. doi: 10.1161/CIRCULATIONAHA.125.076616. Epub 2025 Aug 29. PMID 40884047
- [Derived] Mecinaj A, Gulati G, Heck SL, Holte E, Fagerland MW, Larsen AI, Blix ES, Geisler J, Wethal T, Omland T. Rationale and design of the PRevention of cArdiac Dysfunction during Adjuvant breast cancer therapy (PRADA II) trial: a randomized, placebo-controlled, multicenter trial. Cardiooncology. 2021 Sep 27;7(1):33. doi: 10.1186/s40959-021-00115-w. PMID 34579775

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT03760588/SAP_000.pdf